CLINICAL TRIAL: NCT01583036
Title: An Interaction Study to Assess the Effect of the Ezogabine/Retigabine and the Main Metabolite NAMR on the Pharmacokinetics of Digoxin in Healthy Volunteers
Brief Title: An Open-label, Single-centre Study Evaluating the Pharmacokinetics of Digoxin Alone and When Administered at Various Doses of Ezogabine/Retigabine in Healthy Adults. The Pharmacokinetics of Ezogabine/Retigabine and the N-acetyl Metabolite of Ezogabine/Retigabine (NAMR) Will Also be Assessed
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 116216
Record Dates: First submitted 2012-03-15; First posted 2012-04-23 (Estimated); Last update posted 2018-06-19 (Actual); Status verified 2018-06

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy | interventions — Digoxin; ezogabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Session 1 digoxin alone, Session 2 retigabine plus digoxin (Experimental): Session 1: Single administration of digoxin (0.25mg) and PK assessments up to 144hrs post-dose. Session 2: Retigabine up-titration to 1200mg (TDD) with co-administration of digoxin (0.25mg) at 3 doses or retigabine during the up-titration (600mg, 900mg and 1200mg) and PK assessments up to 144hrs post-dose following wach co-administration.
  Interventions: Drug: Digoxin Alone; Drug: Digoxin + Retigabine

INTERVENTIONS:
Drug: Digoxin Alone — Single administration of digoxin 0.25mg
Drug: Digoxin + Retigabine — Increasing doses of retigabine (300mg, 450mg, 600mg, 750mg, 900mg, 1050mg and 1200mg) administered as TID doses over 44 days. Co-administration with digoxin (0.25mg) on days 10, 24 and 38.

SUMMARY:
An interaction study to assess the effect of the ezogabine/retigabine and the main metabolite NAMR on the pharmacokinetics of digoxin in healthy volunteers

DETAILED DESCRIPTION:
This is an open-label, single-centre study to evaluate the pharmacokinetics of single-dose digoxin alone and when administered at various up titration doses of ezogabine/retigabine in healthy adult subjects. The pharmacokinetics of ezogabine/retigabine and the n-acetyl metabolite of ezogabine/retigabine (NAMR) will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between 18 and 65 years of age inclusive, at the time of signing the informed consent.
* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator and the GSK Medical Monitor agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* A female subject is eligible to participate if she is of: Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) greater than 40 MlU/ml and estradiol less than 40 pg/ml (less than 147 pmol/L) is confirmatory]. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the contraception methods in the protocol if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrollment. For most forms of HRT, at least 2-4 weeks should elapse between the cessation of therapy and the blood draw; this interval depends on the type and dosage of HRT. Following confirmation of their post-menopausal status, they can resume use of HRT during the study without use of a contraceptive method; Child-bearing potential and agrees to use one of the contraception methods listed in the protocol for an appropriate period of time (as determined by the product label or investigator) prior to the start of dosing to sufficiently minimize the risk of pregnancy at that point. Female subjects must agree to use contraception until 1 week post-last dose of ezogabine/retigabine.
* Male subjects with female partners of child-bearing potential must agree to use one of the contraception methods listed in the protocol. This criterion must be followed from the time of the first dose of study medication until at least 1 week post-last dose.
* BMI of 18 to 30 kg/m2 and total body weight greater than 50 kg (110 lbs).
* Normal creatinine clearance assessed by the Cockcroft-Gault Method.
* Subject's aspartate aminotransferase, ALT, alkaline phosphatase, and bilirubin are greater than and equal to 1.5 × ULN (isolated bilirubin greater than 1.5 × ULN is acceptable if bilirubin is fractionated and direct bilirubin less than 35%).
* Subject is a nonsmoker (defined as a nonsmoker during the last 3 months prior to Screening and have a negative cotinine test at screening).
* Subject has a negative drug screen (amphetamines, barbiturates, cocaine metabolites, opiates, benzodiazepines, and cannabinoids) at Screening and at check-in at Day -1.
* Subject is capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.

Exclusion Criteria:

* Subject has positive test results for hepatitis B surface antigen, positive hepatitis C virus, or human immunodeficiency virus (HIV)-1 or -2 at Screening
* Has active suicidal plan/intent or has had active suicidal thoughts in the past 6 months. Has history of suicide attempt in the last 2 years or more than 1 lifetime suicide attempt.
* Presence of proteinuria (at least ++) or hematuria or other clinically significant findings in urinalysis at screening.
* Has a history of urinary retention or risk factors for urinary retention that in the Investigator's judgment could potentially affect subject safety.
* Subject has a history of syncope, clinically significant palpitations, bradyarrhythmia or tachyarrhythmia conduction abnormality (e.g., atrioventricular block of any degree, e.g., left bundle-branch block, right bundle-branch block), or Wolf-ParkinsonWhite syndrome, or any clinically relevant abnormality identified on the screening medical assessment, laboratory examination, ECG, or immunogenicity test
* Subject's blood pressure is greater than and equal to 140/90 mm Hg or heart rate is greater than 100 beats/min at Screening; repeat blood pressures should be taken if the subject's blood pressure is greater than and equal to 140/90 mm Hg and if the results are consistently greater than and equal to 140/90 mm Hg, then the subject should be excluded and advised to consult a physician.
* Subject's QTc interval is greater than 450 ms (per ECG machine interpretation) at screening; repeat measurement should be taken if the QTc greater than 450 ms and if the results are consistently greater than 450 ms, then the subject should be excluded
* Female subject is pregnant or breast-feeding
* Subject has a history of any anaphylactic reaction to any drug or a known hypersensitivity to: LANOXIN/digoxin and/or its excipients, or other digoxin-like medications; or Ezogabine/retigabine; History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Subject has a history of significant cardiovascular or pulmonary dysfunction prior to Screening
* Subject has a fasting triglyceride level greater than 300 mg/dL at Screening
* Subject has a current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert syndrome or asymptomatic gallstones)
* Subject has a history of alcohol or substance abuse within the last 2 years
* Subject has donated blood in the excess of 500 mL within 56 days prior to dosing or intention of donating in the month after completing the study
* Subject has a history of gastrointestinal surgery which could influence gastric emptying (e.g., gastrectomy, gastric bypass)
* Subject has a history of inflammatory bowel disease or irritable bowel syndrome
* Subject has received an investigational drug within 30 days prior to dosing with study medication or 5 half-lives, whichever is longer
* Subject is unlikely to comply with the study protocol and/or to complete the study or required study procedures or is unlikely or unable to return for follow-up visits
* Subject has used prescription medications or over-the-counter medications, herbal supplements, or multivitamins within 14 days prior to dosing with any study medication (beginning with the first dose of digoxin) (see Section 9.2 for additional details)
* Subject has consumed grapefruit juice, cranberry products (such as juice, fruit, or nutritional supplements), or alcohol, caffeine , or xanthine-containing products within 7 days (or 5 elimination half lives whichever is shorter) prior to start the dosing with study medication

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-01-16 (Actual); Primary Completion 2012-04-17 (Actual); Study Completion 2012-04-17 (Actual)

PRIMARY OUTCOMES:
Area under the curve of digoxin from zero hours to infinity (Session 1 day 1 & Session 2 days 10, 24 and 38) | 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 18, 24, 48, 72, 96, 120 and 144 hours post dose
CLr (Renal clearance) of digoxin. Session 1 day 1 & Session 2 days 10, 24 and 38 | 0 to 12 hours, 12 to 24 hours, and 24 to 48 hours post dose
CL/F (Apparent clearance following oral dosing) of digoxin/ Session 1 day 1 & Session 2 days 10, 24 and 38 | 0 to 12 hours, 12 to 24 hours, and 24 to 48 hours post dose

SECONDARY OUTCOMES:
Cmax (Maximum observed concentration) of digoxin. Session 1 day 1 & Session 2 days 10, 24 and 38 | pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 18, 24, 48, 72, 96, 120 and 144 hours post dose
Tmax (Time of occurrence of Cmax) of digoxin. Session 1 day 1 & Session 2 days 10, 24 and 38 | pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 18, 24, 48, 72, 96, 120 and 144 hours post dose
T 1/2 (Terminal phase half-life) of digoxin. Session 1 day 1 & Session 2 days 10, 24 and 38 | pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 18, 24, 48, 72, 96, 120 and 144 hours post dose
Area under the curve of digoxin from zero to 48 hours. Session 1 day 1 & Session 2 days 10, 24 and 38 | pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 18, 24, 48, 72, 96, 120 and 144 hours post dose
Area under the curve of digoxin from zero to 144 hours. Session 1 day 1 & Session 2 days 10, 24 and 38 | pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 18, 24, 48, 72, 96, 120 and 144 hours post dose
Ae (Urinary recovery of unchanged drug) of digoxin from zero to 48 hours. Session 1 day 1 & Session 2 days 10, 24 and 38 | 0 to 12 hours, 12 to 24 hours, and 24 to 48 hours post dose
Cmax of NAMR and ezogabine / retigabine. Days 10, 24 and 38 | pre dose, 0.25, 0.5 1, 1.5, 2, 3, 4, 6, and 8, hours post dose.
Tmax of NAMR and ezogabine / retigabine. Days 10, 24 and 38 | pre dose, 0.25, 0.5 1, 1.5, 2, 3, 4, 6, and 8, hours post dose.
Area under the curve of NAMR and ezogabine / retigabine from zero hours to τ (Time of last observed quantifiable concentration). Days 10, 24 and 38 | pre dose, 0.25, 0.5 1, 1.5, 2, 3, 4, 6, and 8, hours post dose.
Safety and Tolerability (AE's, clinical laboratory, vital signs assessments, ECG's and C-SSRs) | Session 1 day 1 to Session 2 follow-up

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Crean C, Tompson D, Buraglio M. Effects of ezogabine/retigabine on the pharmacokinetics of digoxin in healthy volunteers: results from a drug-drug interaction Phase I study . Epilepsia. 2013;54(Suppl. 3):166.
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study 116216 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/116216?search=study&study_ids=116216#rs
- Available data/document: Study Protocol: 116216 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 116216 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 116216 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 116216 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 116216 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 116216 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 116216 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register